CLINICAL TRIAL: NCT02356068
Title: Thromboelastometry as a Tool to Predict Bleeding and Transfusion Requirement During Liver Transplantation
Brief Title: Predictions of Bleeding During Liver Transplantation With Thromboelastometry
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Other Study IDs: there is no sponsor
Record Dates: First submitted 2015-01-24; First posted 2015-02-05 (Estimated); Last update posted 2020-07-24 (Actual); Status verified 2018-02

CONDITIONS: Hemorrhage
Keywords: liver transplantation, rotem, bleeding, transfusion
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- liver transplantation recepient: every patient who had a liver transplantation. 3 blood samples (2.7ml) for the ROTEM analysis
  Interventions: Other: ROTEM analysis

INTERVENTIONS:
Other: ROTEM analysis — 3 blood samples for ROTEM analysis

SUMMARY:
Patients with cirrhosis present complex coagulation defects. Conventional coagulation tests (INR, platelets count) can not predict bleeding or blood product requirements during liver transplantation. Thromboelastometry (TEM)analyser measures the viscoelastic of the whole blood coagulation generation and lysis. TEM results are available more rapidly than conventional tests and give additional information regarding coagulation strengh, platelet function, and fibrinolysis.

DETAILED DESCRIPTION:
Historically, orthotopic liver transplantation (OLT) has been associated with major blood loss and the need for massive blood product transfusion . The cause of bleeding during OLT is multifactorial . The extensive surgical trauma plays a major role in the origin of bleeding. This bleeding can be accelerated by defects of the hemostatic system. Hemostatic defects can be divided into those present before the operation and those originating during the surgery. The latter can be classified according to the 3 main systems of hemostasis: coagulation, platelet function, and fibrinolysis. Hyperfibrinolysis is an important cause of non surgical bleeding during OLT .

A significant decrease in blood loss and blood product requirements has been observed during OLT over the past 10 years . This decrease can be explained by increase experience, improvements in surgical and anesthetic techniques, and a better understanding of the various hemostatic abnormalities encountered during OLT.

More than 10 years ago, Reyle-Hahn and Rossaint and Dupont et al stated that it is not necessary to correct coagulation defects before the anhepatic phase. More recently, some authors have a poor correlation between bleeding and the peripheral indices of coagulation in patients with chronic liver disease . These patients with cirrhosis are investigated by means of conventional tests for coagulation and primary hemostasis such as prothrombin time (INR), activated partial thromboplastin time (aPTT), platelet count, and skin bleeding time. Two important studies have raised serious questions about clinical use of INR in both measuring liver disease prognosis and in estimating bleeding risk thus calling into question many common and traditional clinical practices .

Now, it is cleat that conventional tests of coagulation (INR, platelet count, fibrinogen) are not able to predict blood product transfusion requirements and bleeding during liver transplantation.

A substantial body of evidence suggests that the use of blood products is associated with morbidity and mortality . Because 33% of liver recipients had acquired their liver disease through the transfusion of blood products , it is important to establish strategies aimed at decreasing blood losses and consequently the need for transfusion. The ability to predict intraoperative blood loss and transfusion requirements would be of great help to ensure adequate blood products and to enable appropriate therapy for patients at high risk of bleeding.

The ROTEM (TEM) thromboelastometry analyzer based on throboelastographic principles , measures the viscoelastic properties of whole blood coagulation generation and lysis. The instrument provides important global hemostatic information about the plasma-platelet-leucocyte interaction and clot tensile strength . TEM results are available more rapidly than those from laboratory-based conventional coagulation testing and also provide additional information regarding coagulation strength, platelet function, and fibrinolysis. Kang et al 39 using thromboelastogram (TEG) showed a decrease in red blood cells (RBC) use after the introduction of TEG monitoring.

ROTEM analysis includes plasmatic coagulation and fibrinolytic factors and inhibitors, as well as all circulating blood cells and provides clinically important information about quality of the final blood clot.

The aim of this observational study was to determine if ROTEM parameters were able to predict blood losses and transfusion of RBC during a liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* every patient who had a liver transplantation

Exclusion Criteria:

no

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: every patient who had a liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
bleeding and transfusion | 24 hours
  evaluation of bleeding and transfusion peroperatively and 24 hours post-op.

CONTACTS AND LOCATIONS:
Overall Officials: Luc Massicotte, Doctor, Principal Investigator — CrCHUM
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

REFERENCES:
- [Derived] Carrier FM, Denault AY, Nozza A, Rioux-Masse B, Roy A, Massicotte L. Association between intraoperative rotational thromboelastometry or conventional coagulation tests and bleeding in liver transplantation: an observational exploratory study. Anaesth Crit Care Pain Med. 2020 Dec;39(6):765-770. doi: 10.1016/j.accpm.2020.07.018. Epub 2020 Oct 1. PMID 33011332